CLINICAL TRIAL: NCT06288906
Title: Acute and Subacute Iliofemoral and/or Caval Deep Vein Thrombosis: Evaluation of Mechanical Thrombectomy Systems in a Monocentric, Observational Retrospective and Prospective Study (ASTER Study)
Brief Title: Acute and Subacute Iliofemoral and/or Caval Deep Vein Thrombosis: Evaluation of Mechanical Thrombectomy Systems
Acronym: ASTER
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Baccellieri Domenico, Principal Investigator, IRCCS San Raffaele
Other Study IDs: ASTER Study
Record Dates: First submitted 2024-02-26; First posted 2024-03-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-03

CONDITIONS: Thrombosis, Venous
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Symptomatic deep vein thrombosis (DVT) patients
  Interventions: Other: mechanical thrombectomy of caval and iliofemoral veins

INTERVENTIONS:
Other: mechanical thrombectomy of caval and iliofemoral veins — investigate efficacy, safety of mechanical thrombectomy systems used in symptomatic acute and subacute ileofemoral and caval thrombosis

SUMMARY:
This is a physician-initiated, observational, monocentric, retrospective and prospective Study. The study is intended to assess the feasibility of mechanical thrombectomy of caval and iliofemoral veins according to normal clinical practice in adult patients with symptomatic acute or subacute ileofemoral or caval deep vein thrombosis objectively diagnosed with CT scan imaging.

DETAILED DESCRIPTION:
Subjects with bilateral DVT may be enrolled, so long as the study limb(s) meet inclusion/exclusion criteria, including IVC patency. It is recommended that in a subject with bilateral DVT, central imaging be performed prior to treatment to evaluate the status of the IVC.

All the visits and procedures described will be performed according to the diagnostic and therapeutic assignment required by clinical practice for the patients under study. Therefore, the choice of assigning the patient to the diagnostic and therapeutic procedures deemed most appropriate for each case is completely independent of the study.

Anticoagulation therapy with enoxaparin sodium (1 mg/kg twice a day) shall be initiated at least 48 hours prior to initiation of study treatment. Hemoglobin, INR, and platelet count must be obtained within 24 hours prior to the mechanical thrombectomy procedure in order to confirm eligibility. The access site is determined by the extent of occlusive disease. When treating a single limb at time, access via the popliteal vein is reasonable.

Upon completion of study treatment, the catheter and sheath shall be removed and hemostasis obtained with pressure over the insertion site followed by placement of a pressure dressing. PCB shall remain placed on both legs until hospital discharge. Anticoagulation therapy with weight based enoxaparin sodium shall also be continued through discharge. The following assessments should be performed following the completion of study treatment, according to the normal clinical practice:

* Duplex imaging (within 24 hours of the completion of treatment)
* Laboratory tests (within 24 hours of the completion of treatment)
* Collection of Adverse Events

ELIGIBILITY:
Inclusion Criteria:

All patients admitted in the Unit of Vascular Surgery with proximal DVT (inferior vena cava, and/or iliac vein, and/or common femoral vein, and/or deep femoral vein, and/or femoral vein), according to ESVS guidelines (2022).

Exclusion Criteria:

* Patient treated with thrombolysis drugs within 48 hours prior to the index procedure
* Active bleeding, recent (<3 months) gastrointestinal (GI) bleeding, active peptic ulcer, severe liver dysfunction, and bleeding diathesis
* Impossibility or refusal to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 50 patients (about 10 cases retrospective and 40 cases prospective) with symptomatic acute or subacute ileofemoral or caval deep vein thrombosis objectively diagnosed with CT scan imaging.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-03-30 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Rate of Technical success | end of the surgical procedure
  restore of vein patency with thrombus removal
Number of Participants presenting Bleeding | 72 hours of mechanical thrombectomy treatment
  Freedom from Major Bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jolly MA, Lockhart MM, Shah D, Huff CM, Valenti EA, Phillips JA, Bittar S, Botti CF, Kolluri R, Silver MJ. Outcomes from a tertiary care center using a catheter thrombectomy system for managing acute iliofemoral deep vein thrombosis. J Vasc Surg Venous Lymphat Disord. 2022 Sep;10(5):1044-1050. doi: 10.1016/j.jvsv.2022.04.010. Epub 2022 Jun 9. PMID 35691538
- [Background] Abramowitz S, Bunte MC, Maldonado TS, Skripochnik E, Gandhi S, Mouawad NJ, Mojibian H, Schor J, Dexter DJ; CLOUT study collaborators. Mechanical Thrombectomy vs. Pharmacomechanical Catheter Directed Thrombolysis for the Treatment of Iliofemoral Deep Vein Thrombosis: A Propensity Score Matched Exploratory Analysis of 12 Month Clinical Outcomes. Eur J Vasc Endovasc Surg. 2024 Apr;67(4):644-652. doi: 10.1016/j.ejvs.2023.11.017. Epub 2023 Nov 21. PMID 37981003
- [Background] Shaikh A, Zybulewski A, Paulisin J, Bisharat M, Mouawad NJ, Raskin A, Ichinose E, Abramowitz S, Lindquist J, Azene E, Shah N, Nguyen J, Cockrell J, Khalsa B, Khetarpaul V, Murrey DA Jr, Veerina K, Skripochnik E, Maldonado TS, Bunte MC, Annambhotla S, Schor J, Kado H, Mojibian H, Dexter D; CLOUT Investigators. Six-Month Outcomes of Mechanical Thrombectomy for Treating Deep Vein Thrombosis: Analysis from the 500-Patient CLOUT Registry. Cardiovasc Intervent Radiol. 2023 Nov;46(11):1571-1580. doi: 10.1007/s00270-023-03509-8. Epub 2023 Aug 14. PMID 37580422